CLINICAL TRIAL: NCT02862327
Title: Intravenous Dexamethasone Versus Placebo for Ultrasound Guided Axillary Brachial Plexus Block With Ropivacaine: Randomised, Controlled, Clinical Trial
Brief Title: Intravenous Dexamethasone for Ropivacaine Axillary Block
Acronym: ADEXA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P/2015/275
Record Dates: First submitted 2016-07-22; First posted 2016-08-11 (Estimated); Last update posted 2018-01-31 (Actual); Status verified 2017-10

CONDITIONS: Postoperative Pain; Anesthesia; Forearm Injuries
Keywords: anaesthetic techniques; regional anesthesia; brachial plexus block; Local Anesthetic; ropivacaine; analgesia; steroid; dexamethasone; placebo; adjuvant; ultrasound guided
MeSH Terms: conditions — Pain, Postoperative; Forearm Injuries; Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- intravenous dexamethasone (Active Comparator): intravenous injection of 8mg (2ml) of dexamethasone during regional anesthesia
  Interventions: Drug: intravenous dexamethasone; Drug: perineural ropivacaine; Other: ultrasound guidance
- intravenous placebo (Placebo Comparator): intravenous injection of 2ml of NaCl 0.9% during regional anesthesia
  Interventions: Drug: intravenous placebo; Drug: perineural ropivacaine; Other: ultrasound guidance

INTERVENTIONS:
Drug: intravenous dexamethasone — intravenous injection of dexamethasone
  Other Names: DEXAMETHASONE MYLAN code UCD 9223084 3400892230849
  Arms: intravenous dexamethasone
Drug: intravenous placebo — intravenous injection of placebo
  Arms: intravenous placebo
Drug: perineural ropivacaine — brachial plexus block with perineural injection of Ropivacaine in the axillary fossa
Other: ultrasound guidance — ultrasound guidance for brachial plexus block in the axillary fossa

SUMMARY:
Prospective monocentric double-blind controlled randomised trial Aim is to assess prolonged postsurgical analgesia by intravenous dexamethasone versus intravenous placebo, after ultrasound guided axillary brachial plexus block

ELIGIBILITY:
Inclusion Criteria:

* ASA 1,2 et 3
* surgery under axillary brachial plexus block
* aged >18 years
* signed information consent

Exclusion Criteria:

* impaired coagulation
* contraindication to regional anesthesia or technical impossibility
* opioids or pain killers abuse or addiction
* steroids consumption in the past 6 months
* dementia or under administrative supervision
* delay of surgery to short to allow regional anesthesia
* pregnancy and breastfeeding
* allergy and contraindication to dexamethasone or ropivacaine
* anticipated bad observation of treatment
* patient enrolled in another trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2017-03-16 (Actual); Study Completion 2017-09-16 (Actual)

PRIMARY OUTCOMES:
Analgesia duration after axillary brachial plexus block | time to first pain at surgical site, an average of 24 hours

SECONDARY OUTCOMES:
Motor block duration after axillary brachial plexus block Safety | up to block recovery, an average of 24 hours
Sensory block duration after axillary brachial plexus block | up to block recovery, an average of 24 hours
incidence of adverse event | 6 month

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Besancon, Besançon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Clement JC, Besch G, Puyraveau M, Grelet T, Ferreira D, Vettoretti L, Pili-Floury S, Samain E, Berthier F. Clinical effectiveness of single dose of intravenous dexamethasone on the duration of ropivacaine axillary brachial plexus block: the randomized placebo-controlled ADEXA trial. Reg Anesth Pain Med. 2019 Mar;44(3):e100035. doi: 10.1136/rapm-2018-100035. PMID 30777900